CLINICAL TRIAL: NCT07334340
Title: Modified vs Standard Crohn´s Disease Exclusion Diet: Evaluation of a Nordic Adaptation of Nutritional Therapy in Paediatric Crohn's Diseas
Brief Title: Modified vs Standard CDED: Evaluation of a Nordic Adaptation of Nutritional Therapy in Paediatric Crohn's Disease
Acronym: N-CDED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Skane University Hospital (Other); Sahlgrenska University Hospital (Other); Göteborg University (Other); Skaraborg Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-05123-01; 282814 (Other Grant/Funding Number: Research and Development Council Fund, Skaraborg Hospital Skövde)
Record Dates: First submitted 2025-12-08; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Pediatric Crohns Disease
Keywords: Pediatric gastroenterology; Crohn´s Disease; Enteral nutrition; Nutritional therapy; whole food; nordic CDED; CDED
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nordic Crohn´s Disease Exclusion Diet (Experimental): 2 weeks of total enteral nutrition followed by 3 phases (6 weeks each) of a Nordic Crohn´s Disease Exclusion Diet.
  Interventions: Other: Nordic Crohn´s Disease Exclusion Diet

INTERVENTIONS:
Other: Nordic Crohn´s Disease Exclusion Diet — The study consists of 20 weeks of dietary intervention, divided into four phases, followed by a 4-week follow-up period. The intervention begins with a 2-week period of liquid nutrition, after which unprocessed foods are gradually introduced while liquid nutrition is progressively reduced over three consecutive 6-week phases. The diet is specifically designed to exclude pro-inflammatory ingredients and emphasize gut-friendly foods. In the final phase, participants are allowed consume most unprocessed foods, along with up to two meals per week containing products with food additives.
  Other Names: N-CDED; Nordic-CDED

SUMMARY:
The primary aim of this clinical trial is to evaluate the clinical effectiveness of the Nordic Crohn's Disease Exclusion Diet (Nordic CDED) in children with Crohn's disease, measured by remission rates, and to compare these outcomes with those reported for the original CDED in similar pediatric populations and study designs.

The secondary objectives are to assess whether the Nordic CDED can facilitate greater individualization of the diet, improve treatment adherence, and enhance quality of life.

The study seeks to answer the following key questions:

* Does the Nordic CDED achieve the same clinical effectiveness as the original CDED?
* Does the Nordic CDED improve adherence and quality of life in children with Crohn's disease? To address these questions, researchers will compare outcomes from children following the Nordic CDED with published results from similar studies of the original CDED, as well as with patients who were not treated with a dietary intervention.

Participant Involvement:

* Follow the Nordic CDED for 20 weeks.
* Attend clinic visits at weeks 2, 8, 14, 20, and 24 for checkups and tests.
* Report adherence to the diet through food records.
* Report quality of life at the beginning and end of the study

DETAILED DESCRIPTION:
The aim of this study is to investigate whether a Nordic version of the Crohn's Disease Exclusion Diet (Nordic CDED) is as effective in achieving clinical remission as the original version of the diet (CDED), which was developed by Levin A et.al. in 2019.

The primary objective is to compare the clinical effect - in terms of remission rates - between Nordic CDED and results from studies where the original CDED has been used in similar patient groups with comparable methodology.

The secondary objective is to evaluate if a Nordic adaptation of the CDED may facilitate individualization and improve adherence and quality of life in paediatric patients with Crohn's Disease.

Overview of the field Crohn's Disease (CD) has increased in prevalence worldwide over the past decades, particularly among children and young people. In Northern Europe, the prevalence is among the highest in the world, with approximately 0.13% of the population living with Crohn's disease. This disease not only causes significant personal suffering and reduced quality of life for affected individuals but also leads to increased healthcare costs. Additionally, it has a major impact on patients' dietary habits, social lives, and self-image. Research has not yet fully clarified why CD develops, but it appears to involve a complex interaction between genetic factors, the immune system, gut microbiota, and environmental influences - with diet playing an increasingly important role.

In the 1990s, exclusive enteral nutrition (EEN), consisting of 6-8 weeks on a liquid diet, was shown to induce remission in patients with mild to moderate active CD. While the underlying mechanism of EEN remains unknown, it has been proposed to favourably modulate the gut microbiome, the intestinal barrier function and immunity. In children with mild to moderate CD, EEN remains the first-line treatment recommended by the European Crohn's and Colitis Organization (ECCO), the European Society for Paediatric Gastroenterology, Hepatology and Nutrition (ESPGHAN), and the Swedish national guidelines. Therefore, this remains a common first-line treatment in the Swedish health-care setting.

However, EEN can be difficult to maintain due to issues such as taste fatigue, poor palatability, nausea, bloating, and the social and psychological burden it places on the patient. As a result, EEN is not considered suitable for long-term management, and many families seek dietary therapies that allow children to eat solid foods.

In recent years, advances in basic and clinical research have greatly expanded our understanding of how dietary factors influence the development and progression of CD. Growing evidence indicates that certain dietary components - particularly ultra-processed foods - may contribute to triggering and maintaining intestinal inflammation in CD.

In line with this new knowledge, CDED was developed - a dietary treatment that has demonstrated comparable efficacy to EEN in achieving corticosteroid-free remission. CDED combines partial enteral nutrition (PEN) with carefully selected foods. Unlike EEN, it includes real food, making it easier for patients to adhere to the treatment while maintaining a more normal lifestyle. Research since 2014 has shown that CDED can help reduce inflammation and maintain remission over time, both in children and adults.

CDED was developed to be adaptable across countries and cultures, using simple and internationally accessible foods, but has so far primarily been applied in Western populations. Implementing a diet-based treatment presents significant challenges in different cultural contexts. Factors such as food availability, patient preferences, religious dietary restrictions, the organization of healthcare services, and societal structures - for example, the fact that schools are often responsible for providing children's meals - mean that dietary adjustments are frequently necessary for the treatment to be feasible, acceptable, and safe in practice. To date, published research on experiences with CDED has primarily been conducted in countries such as Israel, Canada, the USA, and Argentina, as well as several European countries including Spain, Ireland, Sweden, Croatia, and Poland, with ongoing studies in, among others, France and the Netherlands. All these studies confirm the effectiveness of the diet, and among the approximately 20 published studies, several report the need for adaptations - primarily related to the availability of enteral nutrition products and unprocessed foods.

Study Purpose The purpose of this study is to evaluate whether a clinical, cultural, and social adaptation of the CDED to Nordic conditions may improve adherence to dietary treatment among children with CD. It is of utmost importance that this adaptation is carried out without compromising the anti-inflammatory principles of the diet. Such an adaptation is expected not only to enhance adherence but also to reduce the negative impact on quality of life and social well-being for the children and families undergoing dietary treatment. With this knowledge, children would have the opportunity to actively influence their health not only during disease flare-ups but also during symptom-free periods. The overarching goal of this nutritional treatment is to improve gut health by excluding pro-inflammatory foods, without restricting the diet more than necessary.

The aim is for a feasible, culturally adapted version of CDED to be incorporated into Swedish and even Scandinavia IBD treatment guidelines, offering patients additional options for diet-based management. This approach also has the potential to reduce reliance on medications, thereby lowering the risk of side effects and decreasing overall healthcare costs.

If the Nordic CDED proves to be clinically equivalent to the original version, it could serve as a model for how dietary treatments can be adapted to different cultural and social contexts. This, in turn, could contribute to improved adherence and thereby greater treatment efficacy for children with CD in other parts of the world as well. The results from this study will contribute to the growing evidence base for dietary treatment in inflammatory bowel disease and support the development of individualized and more sustainable nutritional strategies for this patient group.

Project description Study design: Multicentre, prospective clinical study including historical controls and non-diet treated controls, utilizing a quantitative approach.

Sample Size: This study is designed as a non-inferiority study, assuming no true difference between the standard and new intervention (i.e., 70% remission/improvement in both groups), a total of 60 patients (30 per group) is required to ensure with 90% power that the 95% confidence interval for the difference between groups excludes a clinically significant difference of 35% or more.

Study Sites: Skaraborg Hospital Skövde, Department of Paediatric Medicine, Queen Silvia Children's Hospital, North Älvsborg County Hospital, Southern Älvsborg Hospital and Skåne University Hospital.

Participants: Children aged 6-18 years with newly diagnosed mild to severe Crohn's disease. Recruitment will begin in at the paediatric gastroenterology clinic at Skövde Hospital. From June 2026, the other remaining hospitals will be included in the study to support recruitment and achieve the required sample size.

Intervention Group: children (6-18 years) with newly diagnosed mild to severe Crohn's disease who are candidates for dietary treatment based on the decision by the patient's treating physician.

Historical Control Group (1): Consists of data from previously published studies in which the original CDED has been used in comparable patient groups. These studies should have been conducted with a similar study design, e.g., prospective clinical studies including children with CD treated with CDED, and where clinical remission was used as the primary outcome measure.

Control Group (2): Patients with Crohn's disease who were not treated with dietary therapy and are diagnosed during the project's recruitment period.

Treatment Protocol:

* Phase 0 (weeks 0-2): Exclusive Enteral Nutrition (liquid diet only)
* Phase 1 (weeks 3-8): Combines partial enteral nutrition (PEN) using an enteral formula with a limited selection of permitted foods, while excluding processed foods, animal fats, gluten, dairy, and other pro-inflammatory or microbiota-disrupting components.

The proportion of PEN will be determined by the research dietitian based on the patient's nutritional status. In cases of acute malnutrition, defined as a BMI < -2 SD, or evidence of linear growth deceleration indicative of chronic undernutrition, the patient will initiate the CDED with 50% of their daily energy requirements provided through PEN. Patients with a normal nutritional status will receive 25% of their daily energy requirements from PEN.

• Phase 2 (weeks 9-14): Gradual reintroduction of additional whole foods and continued exclusion of specific harmful dietary components.

The proportion of PEN will be reduced by 25%; patients who initiated CDED with 50% PEN will continue with 25%, while those who started with 25% PEN will discontinue PEN altogether.

• Phase 3 (weeks 15-20): Further liberalization of the diet while continuing to avoid identified detrimental foods to support long-term remission and gut health. PEN is discontinued at this stage in all patients.

Enteral Formula (liquid diet):

In line with previously published studies using CDED, the enteral product should have certain characteristics: 1.3-1.5kcal/mL, 35-40% fat, 3,5-5g protein/100mL and no fibre. The products may include maltodextrin, soy lecithin and milk fat. To provide different flavours and consistencies 3 different brands will be chosen.

Nordic CDED The diet includes three categories: recommended, permitted, and not permitted food.

Recommended foods: Foods consumed daily to meet protein needs and increase starch and pectin intake, supporting gut microbiota.

Permitted foods: Unprocessed foods required to ensure nutritional adequacy, including protein-, carbohydrate- and fat-rich foods, fruits, vegetables, herbs, spices and beverages.

Not permitted foods: Primarily ultra-processed foods, red and processed meats, animal fat, protein sources high in taurine, gluten and wheat protein, and food additives (e.g. maltodextrin, emulsifiers, artificial sweeteners, carrageenan and sulphites). Fruits and vegetables high in seeds, insoluble fibre or gas-producing carbohydrates are also limited.

Treatment failure: Failure to achieve PCDAI < 15 at week 8 or any physician-initiated treatment change other than immunomodulators (e.g. biologics or corticosteroids).

Study interruption: In case of unexpected complications or incidental findings, patients will be referred for appropriate care. Discontinuation of dietary treatment and study withdrawal will be decided jointly by the physician, dietitian and nurse.

Complications: Diarrhoea or/and worsening of abdominal pain, blood in stool, vomiting, constipation (infrequent defecation, painful defecation, or both).

Data Collection: Data will be collected from medical records and patient-reported outcomes using validated questionnaires. For the controls without nutritional treatment, the information will be taken from SWIBREG register. The REDCap system will be used as the electronic Case Report Form (eCRF).

Measurement Tools:

* Clinical (Week 2, 8, 14, 24): Paediatric Crohn's Disease Activity Index (PCDAI)
* Anthropometric (Week 0, 8, 14, 24): Weight, height, BMI (Z-score)
* Biomarkers (Week 0, 8, 14, 24): C- Reactive Protein (CRP), Erythrocyte Sedimentation Rate (ESR), Albumin (Alb), Faecal Calprotectin (FC)
* Dietary adherence (Week 2, 8, 14, 24): Web-based Food Frequency Questionnaire, 24-hour dietary record and 3-day food diaries.
* Quality of Life (Week 0 and 24): IMPACT III

Evaluation tools:

Food Frequency Questionnaire (SchoolMeal-Q, JuniorMeal-Q and TeenMeal-Q): Validated interactive web-based questionnaires for assessing diet quality.

Modified MARS compliance questionnaire: A questionnaire developed to evaluate compliance to the enteral nutrition and CDED diet.

5-point Likert Scale: A questionnaire developed to evaluate compliance to the diet therapy.

IMPACT III: A valid and reliable questionnaire developed to measure health-related quality of life in Swedish children with inflammatory bowel disease.

Assessment of compliance:

Compliance will be assessed per protocol using three criteria:

1. Treatment continuation: Patients who discontinue the diet due to intolerance or refusal will be classified as having poor compliance.
2. MARS questionnaire: Adherence will be assessed using Question 1 of the modified MARS questionnaire. A response of "always" will be defined as high compliance.
3. Clinical assessment: Compliance will also be evaluated by the physician and dietitian through direct questioning. At week 8, a response of "always" will indicate high compliance; at week 14, "always" or "very often" will indicate high compliance.

High compliance requires fulfilment of all three criteria. Any other response will be classified as poor compliance.

Data analysis and statistics Descriptive data will be presented as median (min-max) for continuous variables and as frequency and percentage for categorical variables.

Comparisons between the intervention group and historical controls will be performed using one-sample tests (Kolmogorov-Smirnov or Wilcoxon signed-rank tests) for numerical variables, and χ² or Fisher's exact tests for categorical variables. Changes over time within the intervention group will be analyzed using Friedman's test.

A p-value ≤ 0.05 will be considered statistically significant. Statistical analyses will be conducted using IBM SPSS Statistics (version 25.0).

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-18 years with recent (<36 months) mild-to-severe CD diagnosis (defined as Paediatric Crohn's Disease Activity Index [PCDAI] 15-47.5)
* Evidence of active inflammation (C-reactive protein [CRP] ≥ 0.5 mg/dL, erythrocyte sedimentation rate [ESR] ≥ 20 mm/h, and/or faecal calprotectin [FCP] ≥ 200 mg/g during screening)
* Stable use of medication other than steroids.

Exclusion Criteria:

* Eating disorders,
* Active extraintestinal manifestations
* Use of systemic corticosteroids
* Active perianal disease
* Positive stool cultures for pathogens, parasites, or Clostridioides difficile
* Fever >38.3°C
* Documented cow's milk protein allergy
* Diabetes, celiac disease and/or psychosocial difficulties.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Corticosteroid-free Clinical Remission | From enrollment to week 8,14 and 24
  Measured by remission rates: PCDAI ≤10 without systemic steroid use, of the Nordic CDED compared to same outcome from studies of the original CDED in similar paediatric populations and study designs.
  Tool: PCDAI, a validated tool used to measure the severity of Crohn's disease in children and adolescents by scoring various clinical and laboratory factors Symptoms: Abdominal pain, frequency/consistency of stools, blood in stool.
  Growth: Weight stability and linear growth (height velocity). Physical Exam: Presence of perianal disease (fistulas, fissures) and extra-intestinal manifestations (arthritis, uveitis, skin issues).
  Lab Tests: Hemoglobin, hematocrit, ESR (Erythrocyte Sedimentation Rate).

SECONDARY OUTCOMES:
Corticosteroid-free clinical remission | At week 8, 14, 20 and 24
  PCDAI < 10
Additional medical treatment | At week 14 of treatment
  Any treatment changed by physician discretion besides immunomodulator (e.g., biologics, steroids).
Reduction in Faecal calprotectin | By week 20 and 24 of the study.
  ≥50% reduction of faecal calprotectin compared to basal concentration.
Adherence to N-CDED diet | Week 2, 8, 14 and 24
  Dietary adherence evaluated by:
  Food Frequency Questionnaire: Validated interactive web-based questionnaires for assessing diet quality.
  24 hour and 3 days food diary recall Modified MARS compliance questionnaire: A questionnaire developed to evaluate compliance to the enteral nutrition and CDED diet.
  5-point Likert Scale: A questionnaire developed to evaluate compliance to the diet therapy.
Modification in quality of life | Basal, week 8 and 24
  Evaluation of the changes in quality of life before, during and after the diet:
  Tool: IMPACT III questionnaire (Inflammatory Bowel Disease Measure for Pediatric, Adolescent, and Children's Thoughts), currently the most widely used, disease-specific instrument for measuring health-related quality of life in children and adolescents with IBD.
  Questions: 35 Rating: From 35 (worst) to 175 (best). Higher total and domain scores consistently indicate better health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Stine Störsrud, RD, PhD, Study Chair — Dept of Molecular & Clinical Medicine, Sahlgrenska Academy, Univ of Gothenburg, Sweden; Elin Malmgren Hård af Segerstad, Ped Diet, PhD, Study Chair — Pediatric Research Institute, Oslo Univ Hosp, Norway; Clinical Sciences, Lund Univ, Malmö, Sweden; Karl Mårild, MD, PhD, Study Director — Dept of Pediatrics, Institute of Clinical Sciences, Sahlgrenska Academy, Gothenburg; Nalleli Vivanco Karlsson, Ped Diet, PhD, Principal Investigator — Dept of Pediatrics, Skaraborg Hosp, Skövde, Sweden; Sahlgrenska Academy, Gothenburg
Locations (3):
- Sweden (3):
  - Skånes University Hospital, Malmo, Skåne County
  - Queen Silvia's Children's and Adolescent Hospital, Gothenburg
  - Skaraborg Hospital Skövde, Pediatric Clinic, Skövde

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to patient privacy concerns and the risk of re-identification, particularly given the small study population.

REFERENCES:
- [Background] Landorf E, Hammond P, Abu-Assi R, Ellison S, Boyle T, Comerford A, Couper R. Formula modifications to the Crohn's disease exclusion diet do not impact therapy success in paediatric Crohn's disease. J Pediatr Gastroenterol Nutr. 2024 Jun;78(6):1279-1286. doi: 10.1002/jpn3.12215. Epub 2024 Apr 16. PMID 38623960
- [Background] Urlep D, Benedik E, Brecelj J, Orel R. Partial enteral nutrition induces clinical and endoscopic remission in active pediatric Crohn's disease: results of a prospective cohort study. Eur J Pediatr. 2020 Mar;179(3):431-438. doi: 10.1007/s00431-019-03520-7. Epub 2019 Nov 28. PMID 31781933
- [Background] Sigall Boneh R, Westoby C, Oseran I, Sarbagili-Shabat C, Albenberg LG, Lionetti P, Manuel Navas-Lopez V, Martin-de-Carpi J, Yanai H, Maharshak N, Van Limbergen J, Wine E. The Crohn's Disease Exclusion Diet: A Comprehensive Review of Evidence, Implementation Strategies, Practical Guidance, and Future Directions. Inflamm Bowel Dis. 2024 Oct 3;30(10):1888-1902. doi: 10.1093/ibd/izad255. PMID 37978895
- [Background] Lijnen P, Petrov V. Transforming growth factor-beta 1-induced collagen production in cultures of cardiac fibroblasts is the result of the appearance of myofibroblasts. Methods Find Exp Clin Pharmacol. 2002 Jul-Aug;24(6):333-44. doi: 10.1358/mf.2002.24.6.693065. PMID 12224439
- [Background] Sigall Boneh R, Park S, Soledad Arcucci M, Herrador-Lopez M, Sarbagili-Shabat C, Kolonimos N, Wierdsma N, Chen M, Hershkovitz E, Wine E, Van Limbergen J. Cultural Perspectives on the Efficacy and Adoption of the Crohn's Disease Exclusion Diet across Diverse Ethnicities: A Case-Based Overview. Nutrients. 2024 Sep 20;16(18):3184. doi: 10.3390/nu16183184. PMID 39339784
- [Background] Sigall Boneh R, Sarbagili Shabat C, Yanai H, Chermesh I, Ben Avraham S, Boaz M, Levine A. Dietary Therapy With the Crohn's Disease Exclusion Diet is a Successful Strategy for Induction of Remission in Children and Adults Failing Biological Therapy. J Crohns Colitis. 2017 Oct 1;11(10):1205-1212. doi: 10.1093/ecco-jcc/jjx071. PMID 28525622
- [Background] Urlep D, Orel R, Kunstek P, Benedik E. Treatment of Active Crohn's Disease in Children Using Partial Enteral Nutrition Combined with a Modified Crohn's Disease Exclusion Diet: A Pilot Prospective Cohort Trial on Clinical and Endoscopic Outcomes. Nutrients. 2023 Nov 4;15(21):4676. doi: 10.3390/nu15214676. PMID 37960328
- [Background] Scarallo L, Banci E, De Blasi A, Paci M, Renzo S, Naldini S, Barp J, Pochesci S, Fioretti L, Pasquini B, Cavalieri D, Lionetti P. A real-life pediatric experience of Crohn's disease exclusion diet at disease onset and in refractory patients. J Pediatr Gastroenterol Nutr. 2024 Sep;79(3):592-601. doi: 10.1002/jpn3.12283. Epub 2024 Jul 4. PMID 38962891
- [Background] Sigall Boneh R, Navas-Lopez VM, Hussey S, Pujol-Muncunill G, Lawrence S, Rolandsdotter H, Otley A, Martin-de-Carpi J, Abramas L, Herrador-Lopez M, Egea Castillo N, Chen M, Hurley M, Wingate K, Olen O, Eurenius Raaf T, Yaakov M, Wierdsma N, Van Limbergen J, Wine E. Modified Crohn's Disease Exclusion Diet Maintains Remission in Pediatric Crohn's Disease: Randomized Controlled Trial. Clin Gastroenterol Hepatol. 2025 Oct;23(11):2001-2011. doi: 10.1016/j.cgh.2024.12.006. Epub 2024 Dec 26. PMID 39732356
- [Background] Sigall-Boneh R, Pfeffer-Gik T, Segal I, Zangen T, Boaz M, Levine A. Partial enteral nutrition with a Crohn's disease exclusion diet is effective for induction of remission in children and young adults with Crohn's disease. Inflamm Bowel Dis. 2014 Aug;20(8):1353-60. doi: 10.1097/MIB.0000000000000110. PMID 24983973
- [Background] Barros VJDS, Severo JS, Mendes PHM, da Silva ACA, de Oliveira KBV, Parente JML, Lima MM, Neto EMM, Aguiar Dos Santos A, Tolentino Bento da Silva M. Effect of dietary interventions on inflammatory biomarkers of inflammatory bowel diseases: A systematic review of clinical trials. Nutrition. 2021 Nov-Dec;91-92:111457. doi: 10.1016/j.nut.2021.111457. Epub 2021 Aug 18. PMID 34583136
- [Background] Roberts I. Safely to school? Lancet. 1996 Jun 15;347(9016):1642. doi: 10.1016/s0140-6736(96)91483-x. No abstract available. PMID 8642954
- [Background] Malmborg P. IBD - Vårdprogram Inflammatorisk tarmsjukdom hos barn och ungdomar (IBD - Care program Inflammatory bowel disease in children and adolescents). In: Svenska Föreningen för Pediatrisk Gastroenterologi HoN-SSAfPG, Hepatology and Nutrition), editor. 2024. p. 21-3.
- [Background] van Rheenen PF, Aloi M, Assa A, Bronsky J, Escher JC, Fagerberg UL, Gasparetto M, Gerasimidis K, Griffiths A, Henderson P, Koletzko S, Kolho KL, Levine A, van Limbergen J, Martin de Carpi FJ, Navas-Lopez VM, Oliva S, de Ridder L, Russell RK, Shouval D, Spinelli A, Turner D, Wilson D, Wine E, Ruemmele FM. The Medical Management of Paediatric Crohn's Disease: an ECCO-ESPGHAN Guideline Update. J Crohns Colitis. 2021 Feb 1;15(2):jjaa161. doi: 10.1093/ecco-jcc/jjaa161. Epub 2020 Oct 7. PMID 33026087
- [Background] Swaminath A, Feathers A, Ananthakrishnan AN, Falzon L, Li Ferry S. Systematic review with meta-analysis: enteral nutrition therapy for the induction of remission in paediatric Crohn's disease. Aliment Pharmacol Ther. 2017 Oct;46(7):645-656. doi: 10.1111/apt.14253. Epub 2017 Aug 16. PMID 28815649
- [Background] de Bie C, Kindermann A, Escher J. Use of exclusive enteral nutrition in paediatric Crohn's disease in The Netherlands. J Crohns Colitis. 2013 May;7(4):263-70. doi: 10.1016/j.crohns.2012.07.001. Epub 2012 Jul 21. PMID 22820027
- [Background] Whelan K, Murrells T, Morgan M, Cummings F, Stansfield C, Todd A, Sebastian S, Lobo A, Lomer MCE, Lindsay JO, Czuber-Dochan W. Food-related quality of life is impaired in inflammatory bowel disease and associated with reduced intake of key nutrients. Am J Clin Nutr. 2021 Apr 6;113(4):832-844. doi: 10.1093/ajcn/nqaa395. PMID 33677550
- [Background] Ng SC, Shi HY, Hamidi N, Underwood FE, Tang W, Benchimol EI, Panaccione R, Ghosh S, Wu JCY, Chan FKL, Sung JJY, Kaplan GG. Worldwide incidence and prevalence of inflammatory bowel disease in the 21st century: a systematic review of population-based studies. Lancet. 2017 Dec 23;390(10114):2769-2778. doi: 10.1016/S0140-6736(17)32448-0. Epub 2017 Oct 16. PMID 29050646
- [Background] Levine A, Wine E, Assa A, Sigall Boneh R, Shaoul R, Kori M, Cohen S, Peleg S, Shamaly H, On A, Millman P, Abramas L, Ziv-Baran T, Grant S, Abitbol G, Dunn KA, Bielawski JP, Van Limbergen J. Crohn's Disease Exclusion Diet Plus Partial Enteral Nutrition Induces Sustained Remission in a Randomized Controlled Trial. Gastroenterology. 2019 Aug;157(2):440-450.e8. doi: 10.1053/j.gastro.2019.04.021. Epub 2019 Jun 4. PMID 31170412

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-09-29): https://cdn.clinicaltrials.gov/large-docs/40/NCT07334340/Prot_SAP_000.pdf
  • Informed Consent Form (2025-09-29): https://cdn.clinicaltrials.gov/large-docs/40/NCT07334340/ICF_001.pdf